CLINICAL TRIAL: NCT01892800
Title: The Pulmonary Vascular / Right Ventricular Response to Lung Resection
Brief Title: Right Side of Heart Function After Lung Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Glasgow (Other)
Collaborators: Golden Jubilee National Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Ben Shelley, Clinical Research Fellow, University of Glasgow
Other Study IDs: 1-shelly
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Lung Cancer; Ventricular Failure, Right
Keywords: Lung Cancer; Ventricular function, Right
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Endo-bronchial aspirate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population - lung resection: Patients with suspected lung cancer undergoing lung resection by anatomic lobectomy
  Interventions: Procedure: Lung resection

INTERVENTIONS:
Procedure: Lung resection
  Other Names: Pulmonary lobectomy

SUMMARY:
The purpose of this study is explore the impact of lung cancer surgery on the function of the right side of the heart.

DETAILED DESCRIPTION:
Lung cancer is the second most common cancer in the UK. In suitable cases the best chance of cure is surgical resection. Studies suggest that lung resection is associated with right ventricular (RV) dysfunction, predisposing to complications and post-operative dyspnoea. Studies of RV function following lung resection have been hampered by the limitations of the techniques used. In addition the mechanism of RV dysfunction has remained elusive.

In this prospective observational study the RV response to lung resection will be characterised by sequential assessment of right ventricular ejection fraction (RVEF) measured using cardiovascular magnetic resonance (CMR). CMR is non-invasive, involves no ionising radiation and due to its high spatial resolution is the gold standard for assessing RV volumes. Comprehensive CMR and echocardiographic assessment of the pulmonary vascular - RV axis will allow us to interpret peri-operative changes in RVEF in the context of RV contractility and loading indices. In addition, contemporaneous blood samples will be taken for measurement of biomarkers of myocardial and endothelial dysfunction and systemic inflammation.

With increased understanding of the mechanisms involved, it may be possible to prevent RV dysfunction; reducing complication rates, hospital stay and costs and ameliorating long term dyspnoea.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Age >16 years
3. Planned elective lung resection by lobectomy

Exclusion Criteria:

1. Pregnancy
2. On-going participation in any investigational research which could undermine the scientific basis of the study
3. Contraindications to magnetic resonance imaging:

   i. Cardiac pacemaker, artificial heart valve, neurostimulator, cochlear implant ii. Aneurysm clips iii. Metal injuries to the eye iv. Loose metal in an part of the body
4. Wedge / segmental / sub-lobar lung resection
5. Pneumonectomy
6. Isolated right middle lobectomy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective observational cohort study in 25 patients presenting for lobectomy for resection of primary lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Right ventricular ejection fraction | 3 days
  The primary objective of this study is determine whether RVEF falls post-operatively in patients undergoing lung resection. The primary outcome is RVEF at 3 days post-lung resection compared to pre-operative values determined by CMR.

SECONDARY OUTCOMES:
Association between RVEF and contractility / loading indices | 3 days
  Changes in RVEF must be interpreted in the context of changes in RV contractility and loading parameters. Changes in pre-load, contractility, afterload, ventriculo-arterial coupling, diastolic function and the position of the mediastinum could all potentially influence RVEF.The following indices will be subject to assessment as secondary endpoints:
  Preload - Right ventricular end-diastolic volume (RVEDV) Contractility - Peak systolic strain and strain rate Afterload - Pulmonary artery (PA) distensibility, PA peak velocitly, PA antegrade flow, Estimated PA systolic pressure,Pulmonary artery acceleration time Ventriculo-arterial coupling: Ea/Emax(CMR) Diastolic function: E/A velocity ratio.
RVEF vs LVEF | 3 days
  Changes in right-sided cardiac function must be interpreted in the context of left-sided function. ΔRVEF will be compared to changes in Left Ventricular Ejection Fraction (LVEF) over the same period.
Association between biomarkers of myocardial and endothelial dysfunction, systemic inflammation, oxidative and nitrosative stress and ΔRVEF | 3 days
  Association between biomarkers of myocardial and endothelial dysfunction, systemic inflammation, oxidative and nitrosative stress and ΔRVEF.
  Myocardial dysfunction: Brain natriuretic peptide and high sensitivity Troponin-T. Systemic inflammation: C-reactive protein and Pentraxin 3. Oxidative / Nitrosative stress: Malondialdehyde, nitrate and nitrite (determined in plasma and endobronchial aspirate and the end of surgery). Endothelial dysfunction:
  Angiopoietin (Ang) 1 & 2, Von Willebrand factor (VWf), E-selectin (ESEL) and soluble intracellular adhesion molecule (sICAM)).
Association between RVEF and functional status | 3 months and 1 year
  Association between RVEFpreop, RVEFpostop, and RVEF3months and functional status by self report and 6-minute walk test (6MWT). Functional status will be assessed subjectively by written questionnaire. Scoring will be based on the New York Heart Association (NYHA) classification, WHO performance status classification and health related quality of life scoring by EQ-5D questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Shelley, MB ChB, Principal Investigator — University of Glasgow
Locations (1):
- Golden Jubilee National Hospital, Clydebank, United Kingdom

REFERENCES:
- [Derived] Glass A, McCall P, Arthur A, Mangion K, Shelley B. Pulmonary artery wave reflection and right ventricular function after lung resection. Br J Anaesth. 2023 Jan;130(1):e128-e136. doi: 10.1016/j.bja.2022.07.052. Epub 2022 Sep 15. PMID 36115714
- [Derived] Young DJ, McCall PJ, Kirk A, Macfie A, Kinsella J, Shelley BG. B-type natriuretic peptide predicts deterioration in functional capacity following lung resection. Interact Cardiovasc Thorac Surg. 2019 Jun 1;28(6):945-952. doi: 10.1093/icvts/ivz016. PMID 30753496